CLINICAL TRIAL: NCT04640012
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics of DC371739 Single-Dose Treatment in Healthy Subjects
Brief Title: Ascending-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics of DC371739 Single-Dose Treatment in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JYD0101
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2022-03

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DC371739 100mg (Experimental): Single dose of 100 mg tablet orally administered
  Interventions: Drug: DC371739
- Placebo (Placebo Comparator): Placebo orally administered
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DC371739 — Participants received one of 6 dose levels of DC371739 administered as single oral doses.
  Arms: DC371739 100mg
Drug: Placebo — Placebo orally administered
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety, tolerability, pharmacokinetics of DC371739 after a single-dose oral administration in healthy Chinese subjects, and to explore the maximum tolerated dose, also the pharmacokinetics of urine and feces.

DETAILED DESCRIPTION:
This is a randomized, double-blind , placebo-controlled, single-dose study in 43 male healthy subjects assigned to one of the six dose groups (30mg、50mg、100mg、 200mg、400mg and 600mg). 30mg dose group is the pilot group with 3 subjects. Each of the other dose groups will include 8 subjects (7 for DC371739 and 1 for placebo). Subjects will be admitted for treatment on day -1 and receive a single dose of study drug or placebo on day 1. Subjects from different dose groups were enrolled in turn, the next dose group was conducted on the premise that the D6 safety evaluation was completed after the administration of the previous dose group with the result was tolerance. Blood samples will be collected for each group after administration for pharmacokinetic data analysis. Urine and feces were collected in three dose groups of 100 mg, 200 mg and 400 mg respectively to explore the pharmacokinetic characteristics of urine and feces.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-40 years, inclusive, male;
2. Weight≥50kg; body mass index of 19 to 26 kg/m2, inclusive;
3. Based on the medical history, physical examination, clinical laboratory examination, 12-lead ECG and vital signs results, subjects with no evidence of active or chronic diseases, or clinically significant abnormalities;

Exclusion Criteria:

1. Subjects with a history of allergy to study drug ingredients or similar drug, with a history of allergic disease or allergic constitution
2. Presence of symptoms or related history of any major disease, including but not limited to heart, liver, kidney diseases or other acute and chronic digestive tract diseases, respiratory diseases, bone and joint diseases, as well as blood, endocrine, nerve, mental and other systemic disease, or any other diseases or physiological conditions that could interfere with the results;
3. Any surgical condition or condition that may significantly affect the metabolism and excretion of drug absorption and distribution, or that may pose a hazard to the subjects participating in the study; Any surgical condition or condition that may significantly affect the absorption, distribution, metabolism, and excretion of the study drug, or any surgical condition or condition that may harm to the subjects participating in the study;
4. Subjects who donated blood or lost 400 ml of blood within 3 months prior to screening;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | From the first dose of study drug until Day 15 in three arms
  The relationship of each adverse event to the investigational product was assessed by the investigator.A serious adverse event (SAE) is defined as an adverse event that is fatal is life threatening (places the subject at immediate risk of death) requires in-patient hospitalization or prolongation of existing hospitalization results in persistent or significant disability/incapacity other significant medical hazard.
Total urine excretion rate | From the first dose of study drug until Day 6
  Urine samples will be taken at different time points for analysis in three arms
Total feces excretion rate | From the first dose of study drug until Day 6
  feces samples will be taken at different time points for analysis in three arms

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC(0-t)) | From the first dose of study drug until Day 6
  Blood samples will be taken at different time points before and after administration.
Time to reach maximum plasma concentration (Tmax) | From the first dose of study drug until Day 6
  Blood samples will be taken at different time points before and after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Song Ai yun, Phd.MD., Study Director — Guang zhou JOYO Pharma
Locations (1):
- Shanghai Xu hui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No